CLINICAL TRIAL: NCT05698563
Title: Clinical Implication of Intermetatarsal Bursitis in Patients With Rheumatoid Arthritis
Brief Title: Intermetatarsal Bursitis in Patients With Rheumatoid Arthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to health-related issues in the research group, that hindered inrolement of patients.
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Danish Rheumatism Association (Other)
Responsible Party: Principal Investigator, Sif Binder Larsen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-22033815
Record Dates: First submitted 2023-01-13; First posted 2023-01-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Intermetatarsal Bursitis; Rheumatoid Arthritis
Keywords: Forefoot pain
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Magnetic Resonance Imaging; Ultrasonography; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: This is a prospective diagnostic study, including a patient and a control group.
  There is a treatment option with standard treatment for the patient group, if there is indication based on the diagnostic imaging.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor is blinded to type of patient they are examining.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient group (Other): Patients with rheumatoid arthritis and forefoot pain.
  Interventions: Diagnostic Test: Magnetic resonance imaging; Diagnostic Test: Ultrasound; Drug: Corticosteroid injection; Other: Clinical foot evaluation; Other: Picture of the feet
- Control group (Other): Patients with other rheumatic diseases and absence of forefoot pain.
  Interventions: Diagnostic Test: Magnetic resonance imaging; Diagnostic Test: Ultrasound; Other: Picture of the feet

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — MRI scan with contrast of the foot or feet
  Other Names: MRI
Diagnostic Test: Ultrasound — Ultrasound scan of the feet
  Other Names: US
Drug: Corticosteroid injection — Administered ultrasound guided to patients with intermetatarsal bursitis
  Arms: Patient group
Other: Clinical foot evaluation — An examination of the feet
  Arms: Patient group
Other: Picture of the feet — To evaluate the presence of V-sign/spreading toes

SUMMARY:
The aim of the study is to investigate the incidence and clinical implications of intermetatarsal bursitis (IMB) in patients with rheumatoid arthritis (RA).

The hypothesis is that IMB is a cause of pain in patients with RA.

DETAILED DESCRIPTION:
Within the recent years more research have focused on IMB in patients with rheumatologic disorders. There is emerging evidence that IMB is an inflammatory alteration in line with synovitis in patients with RA, and presence of IMB have been linked to the early stages of RA, especially due to the focus of the published literature.

The clinical implications of the presence of IMB for the patients are yet to be understood. Limited studies have linked the occurrence of IMB to foot impairment, but no studies have been conducted investigating the direct association between forefoot pain and the presence/absence of IMB.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Forefoot pain and diagnosed with RA (patient group)
* Diagnosed with an axial arthritis (control group)

Exclusion Criteria:

* Age <18 years
* Open wounds or ongoing infection in the forefoot at the time of examination
* Persons with a history of significant trauma in the forefoot, e.g. any fracture or previous surgeries in the forefoot
* Persons who have previously received intermetatarsal treatment (Morton's neuroma or IMB) in the same foot, e.g. injection within 6 months or operation at any time
* Exclusion from MRI scan only:
* Persons with contraindications to participate in MRI scan
* Persons with severely impaired renal function (GFR <30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Incidence of intermetatarsal bursitis on MRI | 8 weeks
  High intensity on T2 weighted images, low signal on T1. Thin peripheral enhancement on T1 contrast enhanced pictures.
Incidence of intermetatarsal bursitis on US | 8 weeks
  Hypoechoic mass between metatarsal heads. Activity on power/color doppler.
Incidence of other pathology on MRI | 8 weeks
  Other than intermetatarsal bursitis
Incidence of other pathology on US | 8 weeks
  Other than intermetatarsal bursitis
Change in Visual Analogue Score (VAS) score | At inclusion, 1 and 3 month(s) post treatment
  Pain score related to the foot pain

SECONDARY OUTCOMES:
Incidence of opening toes | 1 day
  Presence of opening toes/V-sign/spreading toes.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark